CLINICAL TRIAL: NCT05416905
Title: Multicenter Evaluation of Deep Brain Stimulation for Idiopathic Craniofacial Dystonia: Globus Pallidus intErnus or Subthalamic Nucleus
Brief Title: Deep Brain Stimulation for Idiopathic Craniofacial Dystonia: GPi or STN
Acronym: MEIGES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other); Civil Aviation General Hospital (Other); Chinese PLA General Hospital (Other); Beijing Pins Medical Co., Ltd (Industry); Shandong University of Traditional Chinese Medicine (Other); Qilu Hospital of Shandong University (Other); Beijing Fengtai Hospital (Unknown)
Responsible Party: Principal Investigator, Jianguo Zhang, Director of Department of Functional Neurosurgery, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2022022
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Craniofacial Dystonia; Deep Brain Stimulation
Keywords: Craniofacial Dystonia; Deep Brain Stimulation; Globus pallidus internus; Subthalamic nucleus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN-DBS (Experimental): The patients in this group will be treated with STN-DBS.
  Interventions: Device: STN-DBS
- GPi-DBS (Active Comparator): The patients in this group will be treated with GPi-DBS.
  Interventions: Device: GPi-DBS

INTERVENTIONS:
Device: STN-DBS — The patients will be treated with deep brain electrode placement of STN target under local and general anesthesia. Switching the system on: the stimulator will be switched on 3 weeks after surgery to allow time for the brain edema and "stun effect" to wear off. Postoperative medication: The subject taking medication in the past will continue the medication. If the subject with no medication before, will be required not to take medication related to dystonia.
  Other Names: subthalamic necleus-deep brain stimulation
  Arms: STN-DBS
Device: GPi-DBS — The patients will be treated with deep brain electrode implantation of GPi target under local and general anesthesia. Except that the surgical target was GPi, the operation process, stimulator switch-on time, and postoperative medication were the same as those in the STN-DBS group.
  Other Names: globus pallidus internus-deep brain stimulation
  Arms: GPi-DBS

SUMMARY:
MEIGES is a prospective, multicenter, randomized controlled clinical trial with the primary hypothesis that, STN-DBS is non-inferior to GPi-DBS for motor symptoms improvements at 365 days postoperatively in patients with idiopathic craniofacial dystonia.

DETAILED DESCRIPTION:
Evaluating therapeutic effects of GPi-DBS vs. STN-DBS on patients with idiopathic craniofacial dystonia: Clinical data of patients at different treatment time points will be collected, using different clinical assessments. The main purpose is to assess whether STN-DBS is non-inferior to GPi-DBS for motor symptoms improvements at 365 days postoperatively in patients with idiopathic craniofacial dystonia.

Primary endpoints: Differences between the two groups in BFMDRS-M change scores in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS.

Secondary endpoints: Differences between the two groups in BFMDRS-M change scores in the stimulation state from before to 90, 180 days (±14 days) after STN-DBS and GPi-DBS. Differences between the two groups in BFMDRS-D, BDSI, JRS, MMSE, MoCA, HRSD, HAMA, SF-36 and programming parameters change scores in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject (male or female, 18-75 years);
2. Diagnosed with idiopathic craniofacial dystonia for more than 1 year, including at least one of the eye and oromandibular region. Cervical dystonia may be present;
3. Treated with oral drugs or botulinum toxin injections, but with no satisfactory curative effect;
4. Normal cognitive function with MMSE score ≥ 24;
5. Informed consent signed.

Exclusion Criteria:

1. Only cervical dystonia, or combined with dystonia in other parts of the body other than the cervical region;
2. Diagnosed with other neuropsychiatric diseases(Alzheimer's disease, amyotrophic lateral sclerosis, Parkinson's disease, etc.);
3. History of brain surgery;
4. Severe depression with HRSD score ≥ 35;
5. Contraindications to neurosurgery(cerebral infarction, hydrocephalus, cerebral atrophy, sequelae of cerebrovascular disease, etc);
6. Contraindications to CT or MRI scanning(claustrophobia, etc);
7. pregnant or breastfeeding female, or has positive pregnancy test prior to randomization;
8. Contraindications to general anesthesia (severe arrhythmia, severe anemia, abnormal liver and kidney function, etc.);
9. Expected lifetime < 12 months;
10. Currently receiving an investigational drug or device;
11. Other circumstances that the investigator considers unsuitable to participate in this study or that may pose a significant risk to the patient (inability to understand or comply with research procedures and follow-up, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Burke-Fahn-Marsden dystonia rating scale-motor score (BFMDRS-M) difference Day 365 | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Burke-Fahn-Marsden dystonia rating scale-motor score (BFMDRS-M) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. BFMDRS-M contains 4 items of 0-40 and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Burke-Fahn-Marsden dystonia rating scale-motor score (BFMDRS-M) difference Day 90 | 90 days postoperatively compared between groups
  Differences between the two groups in the change of Burke-Fahn-Marsden dystonia rating scale-motor score (BFMDRS-M) in the stimulation state from before to 90 days (±14 days) after STN-DBS and GPi-DBS treatment. BFMDRS-M contains 4 items of 0-40 and higher scores indicate a worse outcome.
Burke-Fahn-Marsden dystonia rating scale-motor score (BFMDRS-M) difference Day 180 | 180 days postoperatively compared between groups]
  Differences between the two groups in the change of Burke-Fahn-Marsden dystonia rating scale-motor score (BFMDRS-M) in the stimulation state from before to 180 days (±14 days) after STN-DBS and GPi-DBS treatment. BFMDRS-M contains 4 items of 0-40 and higher scores indicate a worse outcome.
Burke-Fahn-Marsden dystonia rating scale-disability score (BFMDRS-D) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Burke-Fahn-Marsden dystonia rating scale-disability score (BFMDRS-D) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. BFMDRS-D contains 7 items of 0-30 and higher scores indicate a worse outcome.
Blepharospasm disability index (BDSI) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Blepharospasm disability index (BDSI) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. BDSI contains 6 items of 0-4 (average socre) and higher scores indicate a worse outcome.
Jankovic rating scale (JRS) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Jankovic rating scale (JRS) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. JRS contains 2 items of 0-8 and higher scores indicate a worse outcome.
Mini-mental state examination (MMSE) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of mini-mental state examination (MMSE) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. MMSE contains 30 questions of 0-30 and higher scores indicate a better outcome.
Montreal cognitive assessment (MoCA) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Montreal cognitive assessment (MoCA) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. MoCA contains 8 modules of 0-30 and higher scores indicate a better outcome.
Hamilton depression scale (HRSD) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Hamilton depression scale (HRSD) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. HRSD contains 24 items of 24-77 and higher scores indicate a worse outcome.
Hamilton anxiety scale (HAMA) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of Hamilton anxiety scale (HAMA) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. HAMA contains 14 items of 0-56 and higher scores indicate a worse outcome.
Medical outcomes study shortform-36 (SF-36) difference | 365 days postoperatively compared between groups
  Differences between the two groups in the change of medical outcomes study shortform-36 (SF-36) in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment. SF-36 contains 8 modules of 0-100 and higher scores indicate a better outcome.
Programming parameters difference | 365 days postoperatively compared between groups
  Differences between the two groups in programming parameters change scores in the stimulation state from before to 365 days (±14 days) after STN-DBS and GPi-DBS treatment, including total electrical energy delivered (TEED), contact, voltage, pulse width and frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, MD, PhD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No